CLINICAL TRIAL: NCT06795256
Title: Homework to Help with Stone Dissolution in Retrograde Intrarenal Surgery
Brief Title: Homework in Retrograde Intrarenal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, Bedreddin Kalyenci, Principal Investigator, Adiyaman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HRÜ/24.21.21
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Retrograde Intrarenal Surgery; Stone, Kidney
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Homework to Help with Stone Dissolution in Retrograde Intrarenal Surgery (Experimental)
  Interventions: Behavioral: Percussion and position change in retrograde intrarenal surgery
- Standard Retrograde Intrarenal Surgery (No Intervention)

INTERVENTIONS:
Behavioral: Percussion and position change in retrograde intrarenal surgery — To evaluate the effectiveness of this homework on stone clearance rates after RIRC by giving instructions to the patient in the home environment and suggesting percussion (tapping) and movement/position changes to help spontaneous stone passage.
  Arms: Homework to Help with Stone Dissolution in Retrograde Intrarenal Surgery

SUMMARY:
To evaluate the effectiveness of this homework on stone clearance rates after retrograde intrarenal surgery (RIRS) by instructing the patient in the home environment and suggesting percussion and movement/position changes to assist in spontaneous stone passage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for RIRC

Exclusion Criteria:

* Patients with anatomic abnormalities such as horseshoe kidney, fragments in the calyx diverticulum, infundibular stenosis, pelvi-ureteral junction obstruction or ureteral stenosis.
* Patients with morbid obesity, uncontrolled hypertension, previous cerebrovascular accident, skeletal deformity such as significant coronary artery disease or symptomatic gastro-esophageal reflux disease.
* Patients with lumbar disc herniation who have undergone spinal surgery and are unable to undergo behavioral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
stone free rates | 1 month after the intervention/procedure/surgery

SECONDARY OUTCOMES:
Number of Patients with complications and Number of Patients with need for secondary surgery after retrograde intrarenal surgery | 1 month after the intervention/procedure/surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman University, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR